CLINICAL TRIAL: NCT00153309
Title: Evaluation of the Health Benefits of the People With Arthritis Can Exercise Program
Brief Title: Program Evaluation of People With Arthritis Can Exercise
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Missouri-Columbia (Other); St. Louis University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCCDPHP-0507; CDC-NCCDPHP-MM-0507
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-09

CONDITIONS: Arthritis; Osteoarthritis; Rheumatoid Arthritis
Keywords: arthritis; exercise; physical activity; physical function; pain
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Motor Activity; Pain

INTERVENTIONS:
Behavioral: People with Arthritis Can Exercise

SUMMARY:
The purpose of this study is to evaluate the health and arthritis-specific benefits of participation in the Arthritis Foundation People with Arthritis Can Exercise program and to collect information to improve community-based dissemination of this program.

DETAILED DESCRIPTION:
Only about 24% of people with arthritis report sufficient physical activity to provide general health benefits. Research has demonstrated that many people with arthritis can safely exercise to improve fitness and health. The People with Arthritis Can Exercise (PACE) program, developed by the Arthritis Foundation, is a land-based recreational physical activity and exercise program. PACE has been offered as a community-based program for over 10 years and small studies have reported benefits for people with arthritis. However, there has been no randomized controlled community trials that evaluate the effectiveness of PACE in the community. The goals of the Evaluation of PACE project are to: (1) appropriately evaluate the AF PACE exercise program, and (2) provide information to support effective content, recruitment and programming. Specific objectives for meeting these goals include:

1. Identify the theoretical foundations and constructs for evaluating the program and select and use appropriate outcome measures;
2. Plan and conduct a randomized controlled trial of 8 and 16 week PACE programs;
3. Perform a qualitative evaluation using focus groups of PACE instructors and participants;
4. Disseminate findings and make recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Self-reported arthritis or chronic joint symptoms
* Community-dwelling

Exclusion Criteria:

* Serious medical conditions which would contraindicate exercise
* No severe physical or mental condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2003-06; Study Completion 2005-06

PRIMARY OUTCOMES:
Physical Activity Level - PASE instrument at baseline, 8 and 16 weeks.
Pain Visual Analog Scale - at baseline, 8 and 16 weeks
Physical Function using the Functional Fitness Battery at baseline, 8 and 16 weeks
Self-reported function (HAQ) at baseline, 8 and 16 weeks

SECONDARY OUTCOMES:
Health-related quality of life
Disease status
Self-efficacy for arthritis management
Self-efficacy for exercise
Social support
Depressive symptoms
Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Hootman, PhD, Study Director — Centers for Disease Control and Prevention; Marian Minor, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- St. Louis University, St Louis, Missouri, United States